CLINICAL TRIAL: NCT02016183
Title: ECARD Combination Tablets LD&HD Special Drug Use Surveillance: Long-term Use (12 Months)
Brief Title: Candesartan Cilexetil / Hydrochlorothiazide Combination Tablets Special Drug Use Surveillance: Long-term Use (12 Months)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 220-011; JapicCTI-132362 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2013-12-14; First posted 2013-12-19 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-04

CONDITIONS: Hypertension
Keywords: Drug Therapy
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Candesartan cilexetil / hydrochlorothiazide: Candesartan cilexetil/Hydrochlorothiazide 4 mg/6.25 mg or 8 mg/6.25 mg combination tablets, orally, once daily for up to 12 months. This drug should not be used as a first-line drug for hypertension treatment. Participants received interventions as part of routine medical care.
  Interventions: Drug: Candesartan cilexetil / hydrochlorothiazide

INTERVENTIONS:
Drug: Candesartan cilexetil / hydrochlorothiazide — Candesartan cilexetil / hydrochlorothiazide combination tablets
  Other Names: ECARD® Combination Tablets LD&HD

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of long-term use of candesartan cilexetil / hydrochlorothiazide combination tablets (ECARD) Combination Tablets LD&HD in hypertensive patients in the routine clinical setting

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of candesartan cilexetil / hydrochlorothiazide combination tablets (ECARD combination tablets) to evaluate in hypertensive patients in the routine clinical setting. Because the drug contains a diuretic (hydrochlorothiazide) , it is necessary to assess the safety, especially on serum uric acid. (the planned sample size is 3000).

The usual adult dosage is 1 tablet (4 mg/6.25 mg or 8 mg/6.25 mg as a candesartan cilexetil/hydrochlorothiazide) administered orally once daily. This drug should not be used as a first-line drug for hypertension treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients

Exclusion Criteria:

(1) Patients with a history of hypersensitivity to ingredients of ECARD LD&HD combination tablets, thiazides, or their analogues (e.g. sulphonamide derivatives such as chlortalidone) (2) Patients with anuria or patients under hemodialysis (3) Patients with acute renal failure (4) Patients with noticeably decreased Na and K levels in body fluids (5) Pregnant women or women planning to become pregnant

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 3222 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2012-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 557 investigative sites in Japan, from 01-Apr-2009 to 30-Sep-2012.
Pre-assignment Details: Participants with a diagnosis of hypertension were enrolled to receive candesartan cilexetil/hydrochlorothiazide 4 mg/6.25 mg or 8 mg/6.25 mg combination tablets, orally, once daily for up to 12 months as per routine medical practice.
Groups:
- Candesartan Cilexetil/Hydrochlorothiazide: Candesartan cilexetil/Hydrochlorothiazide 4 mg/6.25 mg or 8 mg/6.25 mg combination tablets, orally, once daily for up to 12 months. This drug should not be used as a first-line drug for hypertension treatment. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Candesartan Cilexetil/Hydrochlorothiazide
Started | 3222
Completed | 3157
Not Completed | 65
Not completed — Case Report Forms Uncollected | 13
Not completed — Protocol Violation | 52

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Candesartan Cilexetil/Hydrochlorothiazide
Number analyzed (Participants) | 3157
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.6 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1746
  Male | 1411
Region of Enrollment [Number; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 3157
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient, inpatient, and outpatient and inpatient (participants who were both outpatient and inpatient during some point at the time and 3 months prior to enrollment).
  Participants
    Outpatient | 3065
    Inpatient | 18
    Inpatient and outpatient | 74
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 24.61 (3.885)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 87.21 (10.458)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 2332
  Current/Ex smoker | 409
  Unknown | 416
Allergy/Predisposition to Hypersensitivity [Count of Participants; unit: Participants]
  Had no Allergy/Predisposition to Hypersensitivity | 2811
  Had Allergy/Predisposition to Hypersensitivity | 345
  Unknown | 1
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had no Medical Complications | 798
    Had Medical Complications | 2359
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had no Medical History | 2603
    Had Medical History | 552
    Unknown | 2
Duration of Disease [Mean (Standard Deviation); unit: Years] | 7.12 (7.289)
Use of Antihypertensive Drug Prior to the Start of the Study Drug [Count of Participants; unit: Participants]
  Had Not Used Antihypertensive Drug | 185
  Had Used Antihypertensive Drug | 2972
Violation of Inclusion or Exclusion Criteria [Count of Participants; unit: Participants]
  Had No Violation | 3154
  Had Any Violation | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Adverse Drug Reactions (ADRs)
Description: ADRs are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Up to 12 months
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan Cilexetil/Hydrochlorothiazide
Number analyzed (Participants) | 3157
Participants | 283

2. Secondary Outcome: Changes From Baseline in Systolic Blood Pressure (SBP) at Each Time Point
Description: Reported data are changes in SBP from baseline at Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, and final assessment.
Time Frame: Baseline, and Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, and Final assessment (up to 12 months)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points. Here 'n' is number of participants analyzed at the given time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil/Hydrochlorothiazide
Number analyzed (Participants) | 3072
mmHg
  Change in SBP at Month 1: number analyzed (Participants) | 2775
  Change in SBP at Month 1 | -13.3 (18.02)
  Change in SBP at Month 2: number analyzed (Participants) | 2516
  Change in SBP at Month 2 | -14.8 (18.48)
  Change in SBP at Month 3: number analyzed (Participants) | 2456
  Change in SBP at Month 3 | -15.4 (19.06)
  Change in SBP at Month 4: number analyzed (Participants) | 2324
  Change in SBP at Month 4 | -15.7 (19.34)
  Change in SBP at Month 5: number analyzed (Participants) | 2205
  Change in SBP at Month 5 | -15.6 (19.17)
  Change in SBP at Month 6: number analyzed (Participants) | 2240
  Change in SBP at Month 6 | -16.1 (18.94)
  Change in SBP at Month 7: number analyzed (Participants) | 2146
  Change in SBP at Month 7 | -15.8 (19.27)
  Change in SBP at Month 8: number analyzed (Participants) | 2071
  Change in SBP at Month 8 | -15.8 (19.12)
  Change in SBP at Month 9: number analyzed (Participants) | 2006
  Change in SBP at Month 9 | -16.4 (18.86)
  Change in SBP at Month 10: number analyzed (Participants) | 1996
  Change in SBP at Month 10 | -16.6 (18.60)
  Change in SBP at Month 11: number analyzed (Participants) | 1903
  Change in SBP at Month 11 | -17.0 (18.88)
  Change in SBP at Month 12: number analyzed (Participants) | 1818
  Change in SBP at Month 12 | -18.1 (18.86)
  Change in SBP at Final | -17.5 (19.87)

3. Secondary Outcome: Changes From Baseline in Diastolic Blood Pressure (DBP) at Each Time Point
Description: Reported data are changes in DBP from baseline at Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, and final assessment.
Time Frame: Baseline, and Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, and Final assessment (up to 12 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil/Hydrochlorothiazide
Number analyzed (Participants) | 3072
mmHg
  Change in DBP at Month 1: number analyzed (Participants) | 2775
  Change in DBP at Month 1 | -6.5 (11.40)
  Change in DBP at Month 2: number analyzed (Participants) | 2516
  Change in DBP at Month 2 | -7.3 (11.52)
  Change in DBP at Month 3: number analyzed (Participants) | 2456
  Change in DBP at Month 3 | -7.6 (11.93)
  Change in DBP at Month 4: number analyzed (Participants) | 2324
  Change in DBP at Month 4 | -7.8 (11.97)
  Change in DBP at Month 5: number analyzed (Participants) | 2205
  Change in DBP at Month 5 | -7.8 (12.01)
  Change in DBP at Month 6: number analyzed (Participants) | 2240
  Change in DBP at Month 6 | -8.0 (12.12)
  Change in DBP at Month 7: number analyzed (Participants) | 2146
  Change in DBP at Month 7 | -8.1 (12.42)
  Change in DBP at Month 8: number analyzed (Participants) | 2071
  Change in DBP at Month 8 | -8.2 (12.32)
  Change in DBP at Month 9: number analyzed (Participants) | 2006
  Change in DBP at Month 9 | -8.5 (12.26)
  Change in DBP at Month 10: number analyzed (Participants) | 1996
  Change in DBP at Month 10 | -8.7 (12.49)
  Change in DBP at Month 11: number analyzed (Participants) | 1903
  Change in DBP at Month 11 | -8.5 (12.37)
  Change in DBP at Month 12: number analyzed (Participants) | 1818
  Change in DBP at Month 12 | -9.1 (12.23)
  Change in DBP at Final | -8.5 (12.59)

4. Secondary Outcome: Changes From Baseline in Pulse Rate at Each Time Point
Description: Reported data are changes in Pulse Rate from baseline at Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, and final assessment.
Time Frame: Baseline, and Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, and Final assessment (up to 12 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minutes
Arm/Group | Candesartan Cilexetil/Hydrochlorothiazide
Number analyzed (Participants) | 2120
Beats per minutes
  Change in Pulse Rate at Month 1: number analyzed (Participants) | 1817
  Change in Pulse Rate at Month 1 | -1.3 (9.16)
  Change in Pulse Rate at Month 2: number analyzed (Participants) | 1667
  Change in Pulse Rate at Month 2 | -1.1 (9.76)
  Change in Pulse Rate at Month 3: number analyzed (Participants) | 1622
  Change in Pulse Rate at Month 3 | -1.3 (9.40)
  Change in Pulse Rate at Month 4: number analyzed (Participants) | 1527
  Change in Pulse Rate at Month 4 | -1.5 (9.91)
  Change in Pulse Rate at Month 5: number analyzed (Participants) | 1464
  Change in Pulse Rate at Month 5 | -1.3 (9.99)
  Change in Pulse Rate at Month 6: number analyzed (Participants) | 1492
  Change in Pulse Rate at Month 6 | -1.5 (10.23)
  Change in Pulse Rate at Month 7: number analyzed (Participants) | 1415
  Change in Pulse Rate at Month 7 | -1.1 (10.45)
  Change in Pulse Rate at Month 8: number analyzed (Participants) | 1370
  Change in Pulse Rate at Month 8 | -1.5 (10.08)
  Change in Pulse Rate at Month 9: number analyzed (Participants) | 1352
  Change in Pulse Rate at Month 9 | -1.6 (10.37)
  Change in Pulse Rate at Month 10: number analyzed (Participants) | 1340
  Change in Pulse Rate at Month 10 | -1.7 (10.58)
  Change in Pulse Rate at Month 11: number analyzed (Participants) | 1278
  Change in Pulse Rate at Month 11 | -1.5 (10.56)
  Change in Pulse Rate at Month 12: number analyzed (Participants) | 1275
  Change in Pulse Rate at Month 12 | -1.8 (10.35)
  Change in Pulse Rate at Final assessment | -1.6 (10.86)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Participants may be represented in more than 1 category.
Arm/Group | Candesartan Cilexetil/Hydrochlorothiazide
Serious Adverse Events (participants affected / at risk) | 72/3157
Other Adverse Events (participants affected / at risk) | 158/3157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan Cilexetil/Hydrochlorothiazide (N=3157)
Bronchopneumonia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pyelonephritis acute (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 1
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 3
Cerebral infarction (Nervous system disorders) | 5
Convulsion (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Cerebral artery stenosis (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 4
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Renal disorder (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Chest discomfort (General disorders) | 2
Death (General disorders) | 2 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Oedema peripheral (General disorders) | 1
Sudden death (General disorders) | 2 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Blood creatinine increased (Investigations) | 2
Blood urea increased (Investigations) | 2
Compression fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 4
Fracture (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan Cilexetil/Hydrochlorothiazide (N=3157)
Hyperuricaemia (Metabolism and nutrition disorders) | 81
Blood uric acid increased (Investigations) | 77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.